CLINICAL TRIAL: NCT07024446
Title: Comparison of Cardiovascular Risks Between Hip Fracture Surgery With Continued （Dual Antiplatelet Therapy ） Within 6 Weeks vs After 6 Weeks Post-（Percutaneous Coronary Intervention）: A Prospective Observational Cohort Study
Brief Title: Comparison of Cardiovascular Risks Between Hip Fracture Surgery With Continued DAPT（Dual Antiplatelet Therapy ） Within 6 Weeks vs After 6 Weeks Post-PCI（Percutaneous Coronary Intervention）: A Prospective Observational Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Continued DAPT after PCI
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: PCI Patients; DAPT(Dual Antiplatelet Therapy); Hip Fracture Surgeries
MeSH Terms: interventions — Zinostatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: Within 6 weeks after PCI
  Interventions: Other: The time interval between PCI and NCS
- Control group: beyond 6 weeks after PCI
  Interventions: Other: The time interval between PCI and NCS

INTERVENTIONS:
Other: The time interval between PCI and NCS — Using 6 weeks post-PCI as the demarcation point, patients within 6 weeks were assigned to the observation group, while those beyond 6 weeks formed the control group.

SUMMARY:
Percutaneous coronary intervention (PCI) is commonly used to treat stable ischemic heart disease. Among patients, 7.5% require surgical treatment, and up to 20% may need noncardiac surgery (NCS) within two years.

Compared to patients without coronary stents, those requiring NCS shortly after PCI face an increased risk of perioperative major adverse cardiac and cerebrovascular events (MACCE), primarily manifested as thrombotic and bleeding events. Guidelines recommend 6-12 months of dual antiplatelet therapy (DAPT) post-PCI to prevent stent thrombosis, which is associated with an elevated risk of perioperative bleeding during NCS. Multiple retrospective studies suggest that the incidence of MACCE decreases as the interval between PCI and NCS lengthens, reaching a risk level similar to non-PCI patients after 12 months. However, other studies indicate that the risk in patients with similar PCI-NCS intervals correlates more with surgical complexity and urgency. Guidelines advise adequate antiplatelet therapy post-PCI to prevent stent thrombosis and recommend avoiding elective surgery within 4-6 weeks after PCI, contingent on bleeding and thrombotic risk assessments.

Many post-PCI patients facing NCS option to delay surgery after weighing the risks of discontinuing antiplatelet therapy versus postponement, which not only reduces quality of life but also increases the risks associated with delayed surgery. Additionally, retrospective studies have found that in unavoidable emergency or time-sensitive surgeries, the heightened perioperative cardiovascular risk is primarily due to the underlying surgical condition affecting organ function, rather than the PCI-NCS interval or antiplatelet therapy discontinuation.

Recent advancements in minimally invasive surgical techniques have reduced trauma and bleeding, leading to broader indications for surgery in patients on anticoagulant or antiplatelet therapy. The widespread use of newer-generation drug-eluting stents (DES) with advanced antiproliferative drugs has further lowered stent thrombosis rates. Moreover, refined PCI techniques minimize vascular injury during stent placement, reducing the likelihood of extra-stent restenosis. From an anesthesiology perspective, concerns for post-PCI surgical patients extend beyond bleeding risks to whether cardiac function can withstand perioperative hemodynamic changes. As surgical and anesthetic techniques evolve, traditional single-method anesthesia is increasingly replaced by combined techniques that ensure adequate analgesia while minimizing hemodynamic disturbances, maintaining oxygen supply-demand balance, and reducing ischemic and bleeding events.

Hip fractures in elderly patients, often termed the "last fracture in life," carry high surgical and anesthetic risks for those with coronary artery disease. While PCI addresses coronary stenosis, the use or discontinuation of antiplatelet therapy exposes patients to bleeding and ischemic risks. The optimal timing for hip fracture surgery is within 48 hours; delays may lead to malunion, prolonged bedrest complications (e.g., pressure sores, pneumonia), and increased deep vein thrombosis risk. Modern hip fracture surgeries (e.g., internal fixation, hip replacement, Proximal femoral nail antirotation internal fixation) are well-established, with reduced bleeding and faster recovery, making it feasible to perform surgery without interrupting antiplatelet therapy.

Existing research primarily consists of retrospective analyses of cardiovascular risk prediction in post-PCI patients undergoing NCS, with no recent prospective studies. Guideline recommendations on PCI-NCS intervals remain unchanged since 2016. Consequently, many PCI patients must delay surgery, enduring unpredictable risks and diminished quality of life.

This study aims to prospectively observe the incidence of MACCE in hip fracture surgery performed within six weeks post-PCI without discontinuing DAPT. The findings may provide evidence for the feasibility of early post-PCI surgery, offer clinicians and patients safer antithrombotic strategies, and present a new option to improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

Normal hs-cTnI levels prior to NCS BMI 20-28 kg/m² Post-PCI procedure, currently on regular DAPT therapy Complete PCI procedural documentation (date, quantity, stent type) Mentally sound, capable of normal communication

Exclusion Criteria:

Abnormal hs-cTnI before NCS; Accompanied by dysfunction of other organs History of other major surgeries Risk factors for stent thrombosis (age >79 years, impaired left ventricular function, stent implantation due to acute coronary syndrome, multiple stents, diabetes, renal insufficiency with creatinine >1.5 mg/dl) Abnormal coagulation function Local anesthesia surgery Inability to cooperate

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease undergoing hip fracture surgery after PCI were divided into two groups: 25 cases in the surgery group within 6 weeks after PCI (observation group) and 25 cases in the surgery group after 6 weeks post-PCI (control group).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative changes in blood High-sensitivity cardiac troponin I （hs-cTnI） levels | From admission to discharge
  Detection using chemiluminescence immunoassay (CLIA)
Electrocardiogram ST-T changes | From admission to discharge
Perioperative surgical site blood loss | Perioperative period
  Including intraoperative blood drainage volume, gauze usage, and postoperative wound bleeding drainage volume
Occurrence of Perioperative Adverse Events and Patient Self-Reported Symptoms | From admission to discharge

SECONDARY OUTCOMES:
Changes in blood hs-cTnI levels | Once a month within six months after discharge.
  Detection using chemiluminescence immunoassay (CLIA)
Electrocardiogram ST-T changes | Once a month within six months after discharge
Occurrence of Perioperative Adverse Events and Patient Self-Reported Symptoms | Half a year after discharge

OTHER OUTCOMES:
Gender | Preoperative
Duration of surgery | postoperative
  Record the time from skin incision initiation to skin suture completion.
PCI Stent Types | Preoperative
  Bare metal stent or drug-eluting stent; if it is a drug-eluting stent, the drug coating used must be recorded.
DAPT treatment status | Preoperative
  Drug names, categories, administration methods, and dosages used in DAPT
Age | Preoperative
Body mass index | Preoperative
  kg/m^2
Other comorbidities | Preoperative
  Such as hypertension, diabetes, cerebrovascular diseases, history of gastrointestinal bleeding, etc.
surgical approach | postoperative
  internal fixation, hip replacement, PFNA（Proximal femoral nail antirotation internal fixation）
Coronary artery stenosis site | Preoperative
  Name of diseased blood vessel in coronary heart disease, myocardial ischemia injury and location